CLINICAL TRIAL: NCT07240064
Title: Erector Spinae Plane Block Versus Modified Thoracoabdominal Nerve Block for Analgesia in Pediatric Laparoscopic Abdominal Surgeries: a Prospective, Randomized Comparative Study
Brief Title: Erector Spinae Plane Block Versus Modified Thoracoabdominal Nerve Block for Analgesia in Pediatric Laparoscopic Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Gbre, doctor mahmoud abdeltawab mahmoud lectrer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-154-2025
Record Dates: First submitted 2025-09-22; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Laparoscopic Abdominal Surgeries; Erector Spinae Plane Block; Modified Thoracoabdominal Nerve Block (M-TAPA)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spinae plane block (Active Comparator)
  Interventions: Procedure: Erector Spinae Plane Block
- Modified thoracoabdominal plane block (Active Comparator)
  Interventions: Procedure: Modified thoracoabdominal plane block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Patients were placed in the lateral decubitus position for block performance. The probe in a sterile sleeve was applied 1-2 cm lateral to the Patients and Methods 44 midline to identify the 11-transverse process by counting upward from the sacrum region. After identifying the erector spinae muscle and transverse processes, a 22- gauge, 50 mm nerve block needle were advanced into the target interfacial plane in the craniocaudal direction using the in-plane technique. After confirming the needle placement, 0.4 ml/kg bupivacaine 0.25% were injected. ESPB was considered successful by the linear spread craniocaudally between the tip of the transverse process and the erector spinae muscle. The same process was repeated for the other side.
  Arms: Erector spinae plane block
Procedure: Modified thoracoabdominal plane block — The patient was positioned in a supine posture. A deep angle was given to the costochondral angle at the edge of the 10th costa with the probe in the sagittal direction to view the lower surface of the costal cartilage in the midline. A 22-G, 50-mm block needle was inserted in the cranial direction using the in-plane technique and the needle tip was moved to the posterior aspect of the 10th costal cartilage. It was noted that the needle tip never crossed the cranial edge of the 10th costal cartilage and 0.4 ml/kg bupivacaine 0.25% were injected into the lower surface of the chondrium. The same process will be repeated for the other side.
  Arms: Modified thoracoabdominal plane block

SUMMARY:
Laparoscopic abdominal surgeries are frequently performed in pediatric patients and are often associated with significant postoperative pain, which, if inadequately managed, may delay recovery and increase the risk of chronic pain. Optimal analgesia is therefore essential. Regional anesthesia techniques have gained prominence for their ability to provide targeted pain relief, reduce systemic analgesic requirements, and improve recovery outcomes. Among these, the MTAPA through the Perichondral Approach (MTAPA) and the ESPB have attracted attention for potential pediatric use. MTAPA, a refinement of the traditional TAPA, targets thoracoabdominal and lower intercostal nerves, offering effective abdominal wall analgesia. Its perichondral approach aims to enhance local anesthetic spread, potentially improving postoperative pain control. ESPB involves depositing local anesthetic between the erector spinae muscle and vertebral transverse processes, producing analgesia through dorsal and ventral rami blockade. Though widely applied in various surgeries, its role in pediatric laparoscopic abdominal procedures is less studied. MTAPA covers a broader dermatomal range than techniques such as the Transversus Abdominis Plane (TAP) or Oblique Subcostal TAP block, particularly for anterior dermatomes, though most adult reports note coverage between T6-T12. Both MTAPA and ESPB have shown promise in adults, yet their comparative efficacy in pediatric laparoscopic abdominal surgeries remains unclear. This study aims to address this knowledge gap. Therefore, this study aimed to compare the effectiveness of the ESPB and the MTAPA in providing postoperative analgesia for pediatric patients undergoing laparoscopic abdominal surgeries. The study was prospective randomized double blinded comparative and was conducted on 50 patients. They were divided into two equal groups: group (A): they received MTAPA block after induction of GA and group (B): they received ESPB after induction of GA. The study will be double blinded in which the patients, and outcome assessors involved will be blinded to the study allocation and outcomes. Patients received GA induction via propofol 1.5-2.5 mg/kg, fentanyl 1 µg/kg and the maintenance dose were sevoflurane 2%, Tracrium 0.03 mg/kg.

DETAILED DESCRIPTION:
This prospective randomized double blinded controlled study was carried out on 50 pediatric patients who scheduled to undergo elective laparoscopic abdominal surgeries admitted to Cairo University Specialized Children Hospital in the duration from …...to…...after the approval of ethical committee. Group M-TAPA (group A) (n=25): Patients received M-TAPA block after induction of GA.

• Group ESPB (group B) (n=25): Patients received ESPB after induction of GA. Patients and outcome assessors were blinded to the group of the patients. A pharmacist who is not involved in the study prepared the interventional medications. Methods

Preoperative assessment:

Medical and surgical history of the patients were taken, clinical examination of the patients was performed and routine laboratory investigations such as CBC, coagulation studies (INR), renal function (serum creatinine) and liver function (SGPT, SGOT) were done. Each patient was instructed about postoperative pain assessment with the Face, Legs, Activity, Cry and Consolability (FLACC) scale. FLACC (0 represents "no pain" while 10 represents "the maximum pain").

Intraoperative:

On entering the operating room: all patients were connected to standard ASA monitoring which included electrocardiography (ECG), non-invasive arterial blood pressure (NIBP) including systolic, diastolic & mean arterial blood pressure (MAP), Oxygen saturation using pulse oximetry. An intravenous wide pore cannula was inserted in the upper limb then preoperative preload in the form of 10 mL/kg of Ringer's lactate solution for 15 minutes were given. General anesthesia (GA) was induced with propofol 1.5-2.5 mg/kg, and fentanyl 1µg/kg. After IV Tracrium 0.15 mg/kg, the endotracheal tube was inserted.

Maintaining GA was done with sevoflurane (2%) and 50% oxygen. Incremental doses of IV Tracrium 0.03mg/Kg will be given. The cases were then mechanically ventilated to sustain end-tidal CO2 levels of 30-35 mmHg. Additional fentanyl bolus dosages of 0.5 µg/kg IV were administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain). ESPB and M-TAPA were performed after the induction of general anesthesia. Both blocks were performed using ultrasound guidance (FUJiFilM sonosite) with a linear probe (6-13 MHz) under complete aseptic conditions. The blocks were administered before the surgical incision, with a waiting period of at least 30 minutes. ESPB and M-TAPA were performed by an experienced anesthesiologist. Aspiration before injection and test dose injection were performed. Both blocks were performed bilaterally to ensure adequate analgesia for both sides of the abdomen. This was essential to achieve full pain relief for laparoscopic abdominal surgeries, which involve multiple abdominal regions.

In (Group A):

The patient was positioned in a supine posture. A deep angle was given to the costochondral angle at the edge of the 10th costa with the probe in the sagittal direction to view the lower surface of the costal cartilage in the midline. A 22-G, 50-mm block needle was inserted in the cranial direction using the in-plane technique and the needle tip was moved to the posterior aspect of the 10th costal cartilage. It was noted that the needle tip never crossed the cranial edge of the 10th costal cartilage and 0.4 ml/kg bupivacaine 0.25% were injected into the lower surface of the chondrium. The same process will be repeated for the other side.

In (Group B):

Patients were placed in the lateral decubitus position for block performance. The probe in a sterile sleeve was applied 1-2 cm lateral to the midline to identify the 11-transverse process by counting upward from the sacrum region. After identifying the erector spinae muscle and transverse processes, a 22- gauge, 50 mm nerve block needle were advanced into the target interfacial plane in the craniocaudal direction using the in-plane technique. After confirming the needle placement, 0.4 ml/kg bupivacaine 0.25% were injected. ESPB was considered successful by the linear spread craniocaudally between the tip of the transverse process and the erector spinae muscle. The same process was repeated for the other side.

Postoperative:

Finally, patients were discharged to post anesthesia care unit (PACU). Postoperative pain was assessed by FLACC score Figure 14. A multi-modal analgesic protocol was used for all patients in all groups in the form IV paracetamol 1gm every 6 hrs. Pain intensity was assessed using the FLACC scale which included categories for Face, Legs, Activity, Cry, and Consolability, rated from 0 (no pain) to 10 (maximum pain) at 0.5, 1, 2, 4, 6, 8, 12, and 24 h postoperatively (87). Rescue analgesia of morphine was given as 0.05 to 0.1 mg/kg bolus if the FLACC scale ≥ 4. The maximum dose of morphine was0.2 mg/kg.

Ethical consideration:

Informed consent was obtained from all parents whose children involved in the study. There were adequate provisions to maintain the privacy of participants and confidentiality of the data are as follows:

* The patients were given the option of not participating in the study if they did not want to.
* We put code numbers to each participant with the name and address kept in a special file.
* We hid the patients' names when we use the research.
* We used the results of the study only in a scientific manner and not to use it in any other aims.

Sample size calculation:

The sample size calculation was done by G*Power 3.1.9.2 (Universitat Kiel, Germany). We performed a pilot study (5 cases in each group), and we found that the mean (± SD) Time to first analgesic was 8.2±3.42h in Group ESPB and 4.6±2.7h in Group M-TAPA. The sample size was based on the following considerations: 1.168 effect size, 95% confidence limit, 95% power of the study, group ratio 1:1, and 4 cases were added to each group to overcome dropout. Therefore, we recruited 25 patients in each group. Statistical analysis Statistical analysis was done by SPSS v26 (IBM Inc., Chicago, IL, USA).Shapiro-Wilks test and histograms were used to evaluate the normality of the distribution of data. Quantitative parametric variables were presented as mean and standard deviation (SD) and compared between the two groups utilizing unpaired Student's t- test. Quantitative non-parametric data were presented as median and interquartile range (IQR) and were analyzed by Mann-Whitney test. Qualitative variables were presented as frequency and percentage and were analyzed utilizing the Chi-square test or Fisher's exact test when appropriate. A two tailed P value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age from 2 to 7 years.

  * Both sexes.
  * American Society of Anesthesiologists (ASA) physical status I and II.
  * Patients undergoing elective laparoscopic abdominal surgeries under general anesthesia.

Exclusion Criteria:

* Known allergies to local anesthetics.

  * Pre-existing chronic pain conditions.
  * Significant hepatic or renal dysfunction.
  * Patients with upper airway infection 2 weeks ago.
  * History of developmental delays, mental retardation, or CNS disease.
  * Congenital spine anomaly.
  * Patients with bleeding and coagulation disorders (e.g., platelet count <100,000/mm³, INR > 1.5).
  * Contraindications to regional anesthesia (

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic request (hours) | 24 hours
  Time to first analgesic request (hours)

SECONDARY OUTCOMES:
Secondary outcome | 24 hours
  Pain score assessed by FLACC score..
  * Hemodynamic Parameters blod pressure in mmhg ,heart rate per mintue.
  * Total intraoperative opioid consumption in ml.
  * Total dose of rescue analgesics within the first 24 hours postoperatively in ml
  * Adverse effects such as hematoma, infection, or signs of local anesthetic
  * toxicity.
  * Degree of parent's satisfaction was assessed on a 5-point Likert scale
  * Incidence of postoperative nausea and vomiting (PONV) weight in kilograms height in meters

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All ipd will be shared
Supporting Information: Study Protocol